CLINICAL TRIAL: NCT06010524
Title: A Retrospective Study of Chronic Hepatitis C Patients Treated With SOF/VEL/VOX: Real Life Study
Brief Title: A Study of Chronic Hepatitis C Patients Treated With SOF/VEL/VOX
Acronym: VOSEVI_Reg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cerrahpasa Medical Faculty Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HEPCTURKEY_2
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; VOSEVI
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, non-interventional study. Investigators from infectious diseases and gastroenterology departments will participate this study.

Patients data will be collected from hospital medical records.

DETAILED DESCRIPTION:
Pangenotypic Sofosbuvir/Velpatasvir/Voxilaprevir for 8-12 weeks has been shown highly effective, safe, and well-tolerated in treating patients with chronic HCV infection in clinical trial settings, however, there are no real-world setting data are available.This is the first opportunity from all over the world to demonstrate SOF/VEL/VOXs efficacy and safety in Real World setting especially for the naive patients.

SOF/VEL/VOX is often positioned in retreatment by international guidelines. Previously the reimbursement guideline in Turkey did not allow patients to be re-treated after the failure of DAA treatments. With current guideline Vosevi is approved as the only option for failures of DAA treatments. In the past years in Turkey, SOF+RBV in GT2, SOF+PEF+RBV in GT3, LDV/SOF in GT1.4-6 patients and Viekirax/Exviera in GT1,4 patients have been used and unfortunately, some patients did not benefit from these suboptimal treatments. The efficacy and safety of SOF/VEL/VOX in patients who have experienced treatment failure in real life will be another objective of the research.

This research will support

1. Efficacy and safety of 8-week Pangenotypic SOF/VEL/VOX for treatment naive non-cirrhotics
2. Efficacy and safety of 12-week Pangenotypic SOF/VEL/VOX for treatment naive compensate cirrhotics
3. Efficacy and safety of 12-week Pangenotypic SOF/VEL/VOX for retreatment of NS5A or NS3A4 and non-NS5A treatment-experienced patients (incl. noncirrhotics and cirrhotics)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as chronic hepatitis C and aged 18 and older
* Patients received SOF/VEL/VOX treatment

Exclusion Criteria:

* Decompensated cirrhotic HCV patients
* Having HCC
* eGFR<30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All CHC patients who received Soforbuvir/Velpatasvir/Voxilaprevir combination therapy will be included in this study. The information of these patients will be recorded retrospectively from the Hospital registry system.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained Virology Response 12 | From start date of treatment to 12 weeks after the completion of treatment
  Rate of the patients with undetectabled HCVRNA after 12 weeks of the completion of SOF/VEL/VOX treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fehmi Tabak, Prof, Principal Investigator — Cerrahpasa Medical Faculty
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No